CLINICAL TRIAL: NCT01575899
Title: Efficacy of Seven-day Combined Rabeprazole Plus Levofloxacin Plus Augmentin for Eradication of Helicobacter Pylori.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early termination due to efficacy
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Ming-Cheh Chen, Principal investigator, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB096-28
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-07

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Levofloxacin; Amoxicillin/clavulanate; Rabeprazole; Eastern Taiwan
MeSH Terms: interventions — Amoxicillin; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levofloxacin-Amoxicillin/clavulanate (Experimental): 7-day levofloxacin, amoxicillin/clavulanate, rabeprazole for Hp eradication.
  Interventions: Drug: Levofloxacin-Amox/clav.
- Clarithromycin-Amoxicillin (Active Comparator): 7-day clarithromycin, amoxicillin, rabeprazole for Hp eradication.
  Interventions: Drug: Clarithromycin-Amoxicillin

INTERVENTIONS:
Drug: Levofloxacin-Amox/clav. — Levofloxacin, 500 mg b.i.d., amoxicillin/clavulanate, 875mg/125mg b.i.d. and rabeprazole, 20 mg b.i.d. for 7 days.
  Other Names: Levofloxacin(Cravit), Amoxicillin/clavulanate(Augmentin) and; Rabeprazole(Pariet) for 7 days.
  Arms: Levofloxacin-Amoxicillin/clavulanate
Drug: Clarithromycin-Amoxicillin — Clarithromycin, 500 mg b.i.d., amoxicillin, 1000 mg b.i.d. and rabeprazole 20 mg b.i.d. for 7 days.
  Other Names: Clarithromycin(Klaricid), Amoxicillin(Hiconcil) and; Rabeprazole(Pariet) for 7 days.
  Arms: Clarithromycin-Amoxicillin

SUMMARY:
This prospective controlled randomized open-label clinical trial is designed to determine the eradication rate of 7-day levofloxacin, amoxicillin/clavulanate and rabeprazole regimen compared with 7-day standard triple therapy for adults infected with Helicobacter pylori in Eastern Taiwan.

DETAILED DESCRIPTION:
BACKGROUND:

The resistance rate of Helicobacter pylori (Hp) to amoxicillin and metronidazole therapy is significantly higher in Eastern Taiwan as compared to national and worldwide rates. The high resistance rate in this territory justified a search for a better eradication regimen for Hp infection.

AIM:

To evaluate the efficacy and tolerability of a combination therapeutic regimen of levofloxacin, amoxicillin/clavulanate and rabeprazole (LAcR) versus a conventional seven-day triple therapy with clarithromycin, amoxicillin and rabeprazole (CAR) for the eradication of Hp infection.

METHODS:

We conducted a open-labeled, prospective, randomized, controlled study in a large tertiary referral hospital in Eastern Taiwan. Hp-positive therapy-naïve patients with a positive CLO test as proven by gastroscopy were recruited for potential random assignment to two 7-day treatment groups: LAcR or CAR (control). The primary end point of this study was to evaluate the eradication rate of LAcR regimen. Hp eradication was assessed using the 13C-urea breath test or CLO test performed at least 4 weeks after end of treatment. Compliance and adverse effects with therapy were determined by phone call or outpatient clinic follow up.

EXPECTED RESULT:

The seven-day LAcR regimen evaluated in this study provided improved Hp eradication efficacy when compared with the traditional seven-day triple therapy in Eastern Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Patient proved with infection of H. pylori in gastric mucosa
* Patient with signed informed consent.

Exclusion Criteria:

* woman in breast feeding or pregnancy.
* allergy or severe adverse effects to drugs used in study.
* severe complications of peptic ulcer disease (like perforation or obstruction).
* patients with history of cancer or failure of major organs.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Cheh CHEN, MD, Principal Investigator — Buddhist Tzu Chi General Hospital
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We included H. pylori-positive adult patients assessed by the rapid urease test and histology during the period December 2007 to December 2009 from the out-patient clinic of a single medical center located at Hualien, Eastern Taiwan.
Pre-assignment Details: We excluded patients under the age of 20, woman in pregnancy or breast feeding, those with concomitant illness or conditions (i.e., cardiopulmonary, hepatic, renal diseases, neoplastic diseases), those with severe complication of peptic ulcer disease, like obstruction or perforation, those with allergy to any of the drugs used.
Groups:
- Levofloxacin-Amox/Clav.: 7-day levofloxacin, amoxicillin/clavulanate, rabeprazole for Hp eradication.
- Levofloxacin-Amox/Clav. (Re-eradication): 7-day levofloxacin, amoxicillin/clavulanate and rabeprazole for re-eradication of patient still with evidence of Hp infection after previous intent of eradication.
Period: Overall Study
Arm/Group | Levofloxacin-Amox/Clav. | Clarithromycin-Amoxicillin | Levofloxacin-Amox/Clav. (Re-eradication)
Started | 73 | 73 | 62 (Included patients still with Hp infection after previous therapy without levofloxacin and Augmentin.)
Completed | 68 | 68 | 60
Not Completed | 5 | 5 | 2
Not completed — Lost to Follow-up | 3 | 4 | 2
Not completed — Protocol Violation | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levofloxacin-Amox/Clav. | Clarithromycin-Amoxicillin | Levofloxacin-Amox/Clav. (Re-eradication) | Total
Number analyzed (Participants) | 73 | 73 | 62 | 208
Age Continuous [Mean (Standard Deviation); unit: years] | 52.82 (12.08) | 54.63 (14.42) | 54.68 (11.81) | 54.01 (12.77)
Age, Customized [Number; unit: participants]
  < 54 years | 38 | 34 | 25 | 97
  >=54 years | 35 | 39 | 37 | 111
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 40 | 38 | 113
  Male | 38 | 33 | 24 | 95
Resident area [Number; unit: participants] — Comparison about resident area of participants, living in urban area or rural area.
  participants
    Urban area | 30 | 24 | 19 | 73
    Rural area | 43 | 49 | 43 | 135
Endoscopic finding [Number; unit: participants] — Comparison between participant's endoscopic finding with or without peptic ulcer disease.
  participants
    With peptic ulcer | 30 | 35 | 21 | 86
    Without peptic ulcer | 43 | 38 | 41 | 122
Follow up method [Number; unit: participants] — Information about the follow up method to confirmed the post-treatment Hp status of participants.
  participants
    C13-UBT | 65 | 65 | 55 | 185
    CLO test | 5 | 4 | 5 | 14
    No follow up | 3 | 4 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Eradication Rate (Participants Naive to Anti-H. Pylori Treatment)
Description: A negative post-treatment 13C-urea breath test or CLO test result at more than 4 weeks after complete use of drug for treatment.
Time Frame: 4 weeks after complete use of drug for treatment
Population: Intent to treat analysis of eradication (negative result of follow up method) measured 4 weeks after complete the treatment, for participants never received anti-H. pylori treatment before.
Measure: Number; unit: percentage of eradicated participants
Arm/Group | Levofloxacin-Amox/Clav. | Clarithromycin-Amoxicillin
Number analyzed (Participants) | 73 | 73
percentage of eradicated participants | 78.1 | 57.5
Statistical Analysis 1: Comparison: Levofloxacin-Amox/Clav. vs Clarithromycin-Amoxicillin; Test type: Superiority or Other; p = 0.008, Chi-squared; Odds Ratio (OR) = 2.629, 95% CI 2-sided [1.28 to 5.42], Standard Error of Mean 3.1526

2. Other Pre Specified Outcome: Re-eradication Rate
Description: Re-eradication successful rate (percentage of participants with a negative result of C13 or CLO test at least four weeks after the 2nd treatment) with 7-day levofloxacin, amoxicillin/clavulanate and rabeprazole for patients still with Hp infection previously treated with regimen without levofloxacin and Augmentin.
Time Frame: 4 weeks after complete use of drug for treatment
Population: This intent-to treat analysis is without control group, including patients still with Hp infection previously treated with regimen without levofloxacin and Augmentin.
Measure: Number; unit: percentage of successful re-eradication
Groups:
- Levofloxacin-Amox/Clav. (Re-eradication): 7-day levofloxacin, amoxicillin/clavulanate and rabeprazole for patients still with Hp infection previously treated with regimen without levofloxacin and Augmentin.
Arm/Group | Levofloxacin-Amox/Clav. (Re-eradication)
Number analyzed (Participants) | 62
percentage of successful re-eradication | 72.6

3. Secondary Outcome: Eradication Rate of Participants Living in Rural Area.
Description: Subgroup analysis on eradication rate (percentage of participants with a negative result of C13 or CLO test at least four weeks after treatment) according to resident area of participants, especially who are living in rural area.
Time Frame: 4 weeks after complete use of drug for treatment
Population: Subgroup analysis (intent-to-treat) on eradication rate of participants who are living in rural area of Taiwan.
Measure: Number; unit: percentage of eradicated participants
Groups:
- Levofloxacin-Amox/Clav.: Participants who are living in rural area and received 7-day levofloxacin, amoxicillin/clavulanate and rabeprazole for Hp eradication.
- Clarithromycin-Amoxicillin: Participants who are living in rural area and received 7-day clarithromycin, amoxicillin and rabeprazole for Hp eradication.
Arm/Group | Levofloxacin-Amox/Clav. | Clarithromycin-Amoxicillin
Number analyzed (Participants) | 43 | 49
percentage of eradicated participants | 81.4 | 51.3
Statistical Analysis 1: Comparison: Levofloxacin-Amox/Clav. vs Clarithromycin-Amoxicillin; Test type: Superiority or Other; p = 0.004, Chi-squared; Odds Ratio (OR) = 3.87, 95% CI 2-sided [1.5 to 10.02], Standard Error of Mean 3.2589

ADVERSE EVENTS:
Time Frame: Since participants enrolled into the study till completed the follow up, at least five weeks.
Arm/Group | Levofloxacin-Amox/Clav. | Clarithromycin-Amoxicillin | Levofloxacin-Amox/Clav. (Re-eradication)
Serious Adverse Events (participants affected / at risk) | 1/73 | 0/73 | 0/62
Other Adverse Events (participants affected / at risk) | 10/73 | 11/73 | 17/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Levofloxacin-Amox/Clav. (N=73) | Clarithromycin-Amoxicillin (N=73) | Levofloxacin-Amox/Clav. (Re-eradication) (N=62)
Visited our emergency room (Gastrointestinal disorders) | 1/10 (1) | 0/11 (0) | 0/17 (0) — Vomiting during eradication, visited our ER, improved after symptomatic treatment, then the case was loss in follow up.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levofloxacin-Amox/Clav. (N=73) | Clarithromycin-Amoxicillin (N=73) | Levofloxacin-Amox/Clav. (Re-eradication) (N=62)
Nausea / Hiccough (Gastrointestinal disorders) | 4 (4) | 4 (4) | 4 (4) — Hiccough and/or sensation of nausea
Loose stool / Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 8 (8) — Diarrhea or loose stool passage.
Change in appetite / Bitter sensation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) — Bitter sensation in tongue, change in taste or appetite.
Abdominal fullness / Flatus (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4) — Flatus, abdominal fullness and gas passage.
Insomnia (General disorders) | 1 (1) | 0 (0) | 4 (4) — Poor sleep.

LIMITATIONS AND CAVEATS:
The limitation of this study is the local primary resistance of Hp to levofloxacin and to amoxicillin/clavulanate is unknown. We are currently engaged in an on-going investigation of the influence of CYP2C19 genotypes on this new regimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No